CLINICAL TRIAL: NCT00195611
Title: Observational Study of the Rhinopharyngeal Carriage of Streptococcus Pneumoniae (Sp) in Infants With Acute Otitis Media (AOM)
Brief Title: Study of Streptococcus Pneumoniae in Nose and Throats of Infants With Acute Otitis Media
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Other Study IDs: 0887X-100918
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Otitis Media; Otitis Media With Effusion; Pneumococcal Infections
Keywords: Middle Ear Infection
MeSH Terms: conditions — Otitis Media; Otitis Media with Effusion; Pneumococcal Infections | interventions — Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Drug: Prevenar

SUMMARY:
The aim of this study is to assess in France the impact of Prevenar on the possible evolution of the pneumococcal serotypes distribution and antibiotic resistance in NP samples of children with AOM.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged from 6 to 24 months
* Presenting with AOM (ear infection)
* Patients must not have received any antibiotic therapy within the past 7 days.

Other inclusion applies.

Exclusion Criteria:

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Screening, Cross-Sectional, Defined Population, Prospective Study
Sampling Method: Probability Sample
Enrollment: 3293 (Actual)
Dates: Start 2005-09; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (31):
- France (31):
  - Auch
  - Brest
  - Canne La Boca
  - Chambéry
  - Châlons-en-Champagne
  - Combs-la-Ville
  - Créteil
  - Draguignan
  - Essey-lès-Nancy
  - Fontenay-sous-Bois
  - Grenoble
  - Grigny
  - Lagny
  - Les Lilas
  - Les Ulis
  - Lyon
  - Marquette-lez-Lille
  - Marseille
  - Massy
  - Molsheim
  - Paris
  - Rouen
  - Saint-Brieuc
  - Saint-Maur-des-Fossés
  - Sélestat
  - Thionville
  - Toulouse
  - Tours
  - Vandœuvre-lès-Nancy
  - Vence
  - Villeneuve-lès-Avignon